CLINICAL TRIAL: NCT03116048
Title: Evaluation of Persistent Postsurgical Pain After Breast Surgery With a Pectoral Nerves Block (Pecs) Type II: a Prospective Follow-up After a Prospective Double Blind Placebo-controlled Randomized Controlled Trail
Brief Title: Evaluation of Persistent Postsurgical Pain After Breast Surgery With a Pectoral Nerves Block (Pecs) Type II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GZA Ziekenhuizen Campus Sint-Augustinus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: GZA-ANE-PECS-02
Record Dates: First submitted 2017-04-03; First posted 2017-04-14 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-02

CONDITIONS: Chronic Post-Procedural Pain; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecs group (study group) (Other): Chronic pain assessment with study questionnaire
  Interventions: Other: Chronic pain evaluation
- Control group (placebo group) (Other): Chronic pain assessment with study questionnaire
  Interventions: Other: Chronic pain evaluation

INTERVENTIONS:
Other: Chronic pain evaluation — Chronic pain assessment with study questionnaire

SUMMARY:
Background and objectives The Pectoral Nerves Block (Pecs) Type II is a regional anesthesia technique that provides post-surgical pain relief for patients undergoing breast surgery. Post-procedural pain relief is known to diminish persistent pain. In this prospective follow-up, the investigators evaluated whether the Pecs II block, compared to placebo, is effective in reducing persistent post-procedural pain after breast cancer surgery in female patients.

Patients and methods 140 breast cancer stage 1-3 patients undergoing mastectomy or tumorectomy with sentinel node or axillary node dissection under general anesthesia were randomized to receive a Pecs block (levobupivacaine 0.25%) or placebo (saline 0.9%). Patients were invited between 9 and 31 months after surgery to complete a persistent postsurgical pain survey.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women. For breast cancer patients, surgery is the most effective therapeutic intervention. Up to two thirds of female patients undergoing breast cancer surgery develop chronic post-procedural pain. This can be best understood by the fact that chronic post-procedural pain is strongly associated with acute post-procedural pain and that even minimal breast surgery can result in significant post-procedural pain.

Regional anesthesia techniques can improve acute and chronic post-procedural pain outcomes. In the prospective double blind placebo-controlled randomized controlled trial, the investigators found that the pectoral nerves (Pecs) block type II, as described by Blanco et al., provides reliable and effective post-procedural analgesia for patients undergoing breast surgery.

In this prospective follow-up, the investigators evaluate whether the Pecs II block is effective in reducing chronic post-procedural pain in female adult patients undergoing breast cancer surgery compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* participated in the Large-scale Prospective Double-blind Randomized Controlled Trial of Pecs II Block for Breast Surgery (NCT02544282)

Exclusion Criteria:

* patient refusal

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Chronic post- procedural pain evaluation through questionaire | 1-3 years
  Evaluation of the chronic post procedural pain in breast surgery under general anesthesia with a pecs or placebo block

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Van Houwe, MD, Study Director — GZA Ziekenhuizen Campus Sint-Augustinus
Locations (1):
- GZA Sint Augustinus, Wilrijk, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] El-Tamer MB, Ward BM, Schifftner T, Neumayer L, Khuri S, Henderson W. Morbidity and mortality following breast cancer surgery in women: national benchmarks for standards of care. Ann Surg. 2007 May;245(5):665-71. doi: 10.1097/01.sla.0000245833.48399.9a. PMID 17457156
- [Background] Poleshuck EL, Katz J, Andrus CH, Hogan LA, Jung BF, Kulick DI, Dworkin RH. Risk factors for chronic pain following breast cancer surgery: a prospective study. J Pain. 2006 Sep;7(9):626-34. doi: 10.1016/j.jpain.2006.02.007. PMID 16942948
- [Background] Mejdahl MK, Andersen KG, Gartner R, Kroman N, Kehlet H. Persistent pain and sensory disturbances after treatment for breast cancer: six year nationwide follow-up study. BMJ. 2013 Apr 11;346:f1865. doi: 10.1136/bmj.f1865. PMID 23580693
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328
- [Background] Wu CL, Raja SN. Treatment of acute postoperative pain. Lancet. 2011 Jun 25;377(9784):2215-25. doi: 10.1016/S0140-6736(11)60245-6. PMID 21704871
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Dworkin RH, Turk DC, McDermott MP, Peirce-Sandner S, Burke LB, Cowan P, Farrar JT, Hertz S, Raja SN, Rappaport BA, Rauschkolb C, Sampaio C. Interpreting the clinical importance of group differences in chronic pain clinical trials: IMMPACT recommendations. Pain. 2009 Dec;146(3):238-244. doi: 10.1016/j.pain.2009.08.019. PMID 19836888
- [Background] Wijayasinghe N, Andersen KG, Kehlet H. Analgesic and Sensory Effects of the Pecs Local Anesthetic Block in Patients with Persistent Pain after Breast Cancer Surgery: A Pilot Study. Pain Pract. 2017 Feb;17(2):185-191. doi: 10.1111/papr.12423. Epub 2016 Feb 9. PMID 26857336